CLINICAL TRIAL: NCT03823703
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety, Efficacy, and Pharmacokinetics of Miricorilant in Patients With Presumed Nonalcoholic Steatohepatitis (NASH)
Brief Title: Study Evaluating the Safety, Efficacy, and Pharmacokinetics of Miricorilant in Participants With Presumed Nonalcoholic Steatohepatitis (NASH)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Suspended by sponsor, pending investigation of abnormal laboratory values in patients with NASH
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CORT118335-860
Record Dates: First submitted 2019-01-14; First posted 2019-01-30 (Actual); Results first posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2021-04

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
Keywords: Nonalcoholic Steatohepatitis; NASH; Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — CORT118335

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Miricorilant- 900 mg (Experimental): Participants received 900 mg miricorilant (6 miricorilant tablets of 150 mg) orally once daily.
  Interventions: Drug: Miricorilant
- Miricorilant- 600 mg (Experimental): Participants received 600 mg miricorilant (4 miricorilant tablets of 150 mg and 2 placebo tablets) orally once daily.
  Interventions: Drug: Miricorilant; Drug: Placebo
- Placebo (Placebo Comparator): Participants received 6 placebo tablets orally once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Miricorilant — Tablets taken orally
  Other Names: CORT118335
  Arms: Miricorilant- 600 mg; Miricorilant- 900 mg
Drug: Placebo — Placebo tablets
  Arms: Miricorilant- 600 mg; Placebo

SUMMARY:
This phase 2, double blind, placebo-controlled, randomized study is to assess the safety and efficacy of miricorilant (CORT118335) in patients with presumed Nonalcoholic Steatohepatitis (NASH).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study that assessed the safety efficacy and pharmacokinetics (PK) of miricorilant in patients with presumed Nonalcoholic Steatohepatitis (NASH). Patients who meet the criteria for Study CORT118335-860 were randomized on Day 1 to receive 900 mg miricorilant, 600 mg miricorilant, or placebo for 12 weeks.

Due to observations related to safety, the study was terminated prior to completion and study objectives, endpoints, and procedures were modified as specified in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of NASH based on a biopsy obtained within the last year OR
* Have a diagnosis of presumed NASH based on blood tests and scans

Exclusion Criteria:

* Have participated in another clinical trial within the last year and received active treatment for NASH
* Have participated in another clinical trial for any other indication within the last 3 months
* Are pregnant or lactating women
* Have a BMI <18 kg/m^2
* Have had liver transplantation or plan to have liver transplantation during the study
* Have type 1 diabetes or poorly controlled type 2 diabetes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director, Study Director — Corcept Therapeutics
Locations (15):
- United States (15):
  - Site 207, Chandler, Arizona
  - Site 208, Glendale, Arizona
  - Site 209, Tucson, Arizona
  - Site 227, Los Angeles, California
  - Site 214, Panorama City, California
  - Site 233, Santa Ana, California
  - Site 234, Port Orange, Florida
  - Site 210, Sarasota, Florida
  - Site 228, Kansas City, Missouri
  - Site 232, East Syracuse, New York
  - Site 211, Austin, Texas
  - Site 213, Edinburg, Texas
  - Site 215, Edinburg, Texas
  - Site 212, San Antonio, Texas
  - Site 226, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twelve adult patients with presumed NASH were enrolled in this study.
Period: Overall Study
Arm/Group | Miricorilant- 900 mg | Miricorilant- 600 mg | Placebo
Started | 3 | 5 | 4
Treated | 3 | 5 | 4
Completed | 0 | 0 | 0
Not Completed | 3 | 5 | 4
Not completed — Sponsor request | 0 | 3 | 4
Not completed — Adverse Event | 3 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Miricorilant- 900 mg | Miricorilant- 600 mg | Placebo | Total
Number analyzed (Participants) | 3 | 5 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (14.74) | 54.2 (19.87) | 43.3 (15.15) | 50.9 (16.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 6
  Male | 1 | 3 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 4
  Not Hispanic or Latino | 1 | 3 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 5 | 3 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 4 | 12
Liver Fat Content (LFC) Assessed by MRI-PDFF [Mean (Standard Deviation); unit: Percentage of liver fat content] | 24.57 (6.038) | 15.70 (6.536) | 19.93 (8.750) | 19.33 (7.526)
Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) & Gamma Glutamyl Transferase (GGT) [Mean (Standard Deviation); unit: Units/Liter (U/L)]
  AST | 35.7 (8.14) | 25.6 (12.76) | 31 (4.08) | 29.9 (9.68)
  ALT | 52.3 (15.63) | 33.2 (15.94) | 54.0 (12.11) | 44.9 (16.86)
  GGT | 52.7 (19.63) | 26.2 (9.20) | 59.0 (50.29) | 43.8 (32.20)
Propeptide of Type III Collagen (Pro-C3) [Mean (Standard Deviation); unit: micrograms/liter (μg/L)] | 16.13 (5.350) | 11.20 (2.189) | 13.73 (4.727) | 13.28 (4.159)
Enhanced Liver Fibrosis Score [Mean (Standard Deviation); unit: ELF score] | 9.713 (1.011) | 9.358 (0.486) | 9.330 (0.805) | 9.438 (0.690)

OUTCOME MEASURES:

1. Primary Outcome: Relative Change From Baseline in Liver Fat Content Assessed by Magnetic Resonance Imaging-Proton Density Fat Fraction
Description: The change from baseline in liver fat content (LFC) by magnetic resonance imaging-proton density fat fraction (MRI-PDFF) for each miricorilant dose level (600 mg, 900 mg) versus placebo was assessed. MRI-PDFF was performed to determine the degree of LFC reduction. The relative change is defined for each participant as %: ([Post-Baseline LFC-Baseline LFC]/Baseline LFC) × 100. Due to observations related to safety, the study was terminated. If the participant had at least 6 weeks of treatment, the assessment was completed at the early termination visit. Due to the small sample size, no formal tests were performed to assess statistical differences between treatment groups.
Time Frame: Baseline and up to ~Day 95
Population: The analysis population included all participants who were randomized to the study and had a post-baseline LFC assessment.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Miricorilant- 900 mg | Miricorilant- 600 mg | Placebo
Number analyzed (Participants) | 3 | 2 | 2
Percent change | -50.28 (13.723) | -22.94 (71.943) | 4.63 (5.232)

2. Secondary Outcome: Number of Participants Achieving a Relative Reduction From Baseline in LFC of ≥30% by MRI-PDFF
Description: The number of participants (defined as responders) with a ≥30% reduction in LFC from baseline by treatment group as assessed by MRI-PDFF. The number of participants with a reduction in LFC from baseline of <30% were defined as non-responders. MRI-PDFF was performed at screening and up to 33 days after last dose of study drug. Due to observations related to safety, the study was terminated. If the participant had at least 6 weeks of treatment, the assessment was completed at the early termination visit. Due to the small sample size, no formal tests were performed to assess statistical differences between treatment groups.
Time Frame: Baseline and up to ~Day 95
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Miricorilant- 900 mg | Miricorilant- 600 mg | Placebo
Number analyzed (Participants) | 3 | 2 | 2
Participants
  Responders with a reduction in LFC from baseline of ≥30% | 3 | 1 | 0
  Non-responders with a reduction in LFC from baseline of <30% | 0 | 1 | 2

3. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase
Description: The change in aspartate aminotransferase (AST) from baseline for each treatment group at the Week 6 visit is summarized. Due to the small sample size, no formal tests were performed to assess statistical differences between treatment groups.
Time Frame: Baseline and Week 6
Population: The analysis population included all participants who were randomized to the study and had a post-baseline AST assessment.
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Miricorilant- 900 mg | Miricorilant- 600 mg | Placebo
Number analyzed (Participants) | 1 | 1 | 2
units per liter (U/L) | 346.0 (NA) — No standard deviation because n=1. | 321.0 (NA) — No standard deviation because n=1. | -9.5 (3.54)

4. Secondary Outcome: Change From Baseline in Alanine Aminotransferase
Description: The change in serum alanine aminotransferase (ALT) from baseline for each treatment group at the Week 6 visit is summarized. Due to the small sample size, no formal tests were performed to assess statistical differences between treatment groups.
Time Frame: Baseline and Week 6
Population: The analysis population included all participants who were randomized to the study and had a post-baseline ALT assessment.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Miricorilant- 900 mg | Miricorilant- 600 mg | Placebo
Number analyzed (Participants) | 1 | 1 | 2
U/L | 810.0 (NA) — No standard deviation because n=1. | 826.0 (NA) — No standard deviation because n=1. | -16 (2.83)

5. Secondary Outcome: Change From Baseline in Gamma-glutamyl Transferase
Description: The change in gamma-glutamyl transferase (GGT) from baseline for each treatment group at the Week 6 visit is summarized. Due to the small sample size, no formal tests were performed to assess statistical differences between treatment groups.
Time Frame: Baseline and Week 6
Population: The analysis population included all participants who were randomized to the study and had a post-baseline GGT assessment.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Miricorilant- 900 mg | Miricorilant- 600 mg | Placebo
Number analyzed (Participants) | 1 | 1 | 2
U/L | 29.0 (NA) — No standard deviation because n=1. | 82.0 (NA) — No standard deviation because n=1. | -26.0 (31.11)

6. Secondary Outcome: Change From Baseline in Propeptide of Type III Collagen
Description: The change in serum propeptide of Type III collagen (pro-C3) from baseline at the Week 6 visit is summarized. Due to the small sample size, no formal tests were performed to assess statistical differences between treatment groups.
Time Frame: Baseline and Week 6
Population: The analysis population included all participants who were randomized to the study and had a post-baseline pro-C3 assessment.
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Miricorilant- 900 mg | Miricorilant- 600 mg | Placebo
Number analyzed (Participants) | 1 | 0 | 2
μg/L | 4.0 (NA) — No standard deviation because n=1. |  | -1.65 (2.475)

7. Secondary Outcome: Change From Baseline in Enhanced Liver Fibrosis Score
Description: The change in enhanced liver fibrosis (ELF) from baseline for each treatment group at the Week 6 visit is summarized. The ELF score combines 3 serum biomarkers (hyaluronic acid, tissue inhibitor of metalloproteinases-1 [TIMP-1] and type III procollagen [PIIINP]) which have been shown to correlate with the degree of liver fibrosis assessed by liver biopsy. Each of these markers is measured by an immunoassay and an ELF score is generated [ELF=2.278+0.851 ln(HA)+0.751 ln(PIIINP)+0.394 ln(TIMP-1)], from which a level of fibrosis severity can be determined; higher ELF scores are associated with worsening liver fibrosis. Due to the small sample size, no formal tests were performed to assess statistical differences between treatment groups.
Time Frame: Baseline and Week 6
Population: The analysis population included all participants who were randomized to the study and had a post-baseline liver fibrosis assessment.
Measure: Mean (Standard Deviation); unit: ELF score
Arm/Group | Miricorilant- 900 mg | Miricorilant- 600 mg | Placebo
Number analyzed (Participants) | 1 | 0 | 2
ELF score | 1.050 (NA) — No standard deviation because n=1. |  | 0.225 (0.459)

8. Other Pre Specified Outcome: Number of Participants With a Relative Reduction in Liver Fat Content ≥50% by Magnetic Resonance Imaging-Proton Density Fat Fraction (MRI-PDFF) for Miricorilant Versus Placebo
Time Frame: Baseline and up to ~Day 95
Measure: Count of Participants; unit: Participants
Arm/Group | Miricorilant- 900 mg | Miricorilant- 600 mg | Placebo
Number analyzed (Participants) | 3 | 2 | 2
Participants
  Responders | 1 | 1 | 0
  Non-Responders | 2 | 1 | 2

9. Other Pre Specified Outcome: Number of Participants With Complete Resolution in Liver Fat by MRI-PDFF for Miricorilant Versus Placebo
Time Frame: Baseline and up to ~Day 95
Measure: Count of Participants; unit: Participants
Arm/Group | Miricorilant- 900 mg | Miricorilant- 600 mg | Placebo
Number analyzed (Participants) | 3 | 2 | 2
Participants
  Responders | 0 | 1 | 0
  Non-Responders | 3 | 1 | 2

ADVERSE EVENTS:
Time Frame: Up to ~Day 95 for all cause mortality, serious adverse events and other non-serious treatment-emergent adverse events (TEAEs) during the study period.
Description: The analysis population included all patients who received at least 1 dose of study medication.
Arm/Group | Miricorilant- 900 mg | Miricorilant- 600 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Miricorilant- 900 mg (N=3) | Miricorilant- 600 mg (N=5) | Placebo (N=4)
Drug-induced liver injury (Hepatobiliary disorders) | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Miricorilant- 900 mg (N=3) | Miricorilant- 600 mg (N=5) | Placebo (N=4)
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 2 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 2 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Due to observations related to safety, the study was terminated by the Sponsor prior to completion. The sample size at the time of study termination did not support formal tests to assess statistical differences between treatment groups, and therefore, no efficacy analyses specified in the protocol were performed. Descriptive statistics for efficacy endpoints are provided, but since no patient reached the Week 12 visit, and therefore, descriptive statistics at Week 12 are not presented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No individual publications will be allowed before publication of the multicenter results, except as agreed with the Sponsor. The Investigator agrees to submit all manuscripts or abstracts to the Sponsor for review before submission to the publisher.

DOCUMENTS (2):
  • Study Protocol (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT03823703/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/03/NCT03823703/SAP_001.pdf